CLINICAL TRIAL: NCT03917485
Title: Bio Metrology of Nonfibrous Mineral Particles in Bronchoalveolar Lavage Fluids
Acronym: REACTIT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: REACTIT; 2018-A00475-50 (Other: ID-RCB)
Record Dates: First submitted 2019-04-04; First posted 2019-04-17 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Occupational Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Broncho-Alveolar Washing Fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of this study is to update the pulmonary retention values of non-fibrous mineral particles in the general population.

This study will provide reference values for the interpretation and diagnosis of the cause of certain respiratory diseases potentially related to mineral particles.

DETAILED DESCRIPTION:
Some non-fibrous mineral particles are responsible for respiratory or systemic diseases, most often of occupational origin. Their use concerns multiple professional sectors.

The bio metrology of these particles, namely their quantification in a biological medium requires reference values. These are essential for clinicians to interpret pulmonary retention in patients who may have been exposed professionally or environmentally to non-fibrous mineral particles.

A comparative study conducted in 2015 by lafp showed an increase in the particulate load of nonfibrous mineral particles, including titanium, in lung parenchyma samples over time.

Bronchoalveolar lavage fluid is typically considered to be representative of the lung for the analysis of nonfibrous mineral particles. The thresholds currently used for the bio metrology of nonfibrous mineral particles in bronchoalveolar lavage fluid samples are based on reference values established more than 20 years ago. It is therefore appropriate to update these reference values by establishing a new control population from the analysis of bronchoalveolar lavage fluid from subjects not exposed to the non-fibrous mineral particles in a professional or environmental manner.

ELIGIBILITY:
Inclusion Criteria:

* Subjects not exposed to Non-fibrous Mineral Particle in a professional and / or environmental way.
* Smokers and non-smokers (or weaners who have been weaned for at least 5 years).
* Acceptance to participate in the protocol.
* Affiliated to a social security scheme.

Exclusion Criteria:

* Suspicion of fibrosing pulmonary pathologies.
* Suspicion of pulmonary sarcoidosis ≥ stage 2, pneumoconiosis.
* Subjects with cystic fibrosis.
* Subjects chronic obstructive pulmonary disease (COPD) stage ≥ 3.
* Presence of serious comorbidities that are life-threatening in the short term.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects not exposed to Non-fibrous Mineral Particle in a professional and / or environmental way
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Number of non fibrous mineral particles in LBA (Bronchoalveolar lavage) (nombre of particles by ml) | 1 month
  Quantitative analysis of Non Fibrous Mineral Particles on samples obtained from subjects selected free from any significant occupational or environmental exposure to Non-fibrous Mineral Particle.

SECONDARY OUTCOMES:
Name of non fibrous mineral particles in LBA (Bronchoalveolar lavage) (nombre of particules by ml) | 1 month
  Identification of particles
seize of non fibrous mineral particles in LBA (Bronchoalveolar lavage) | 1 month
  seize of particles

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No